CLINICAL TRIAL: NCT06025500
Title: Analysing cEllular Bioenergetics aNd Structural aDaptations in the qUadriceps Muscle befoRe and After endobroNChial Valve treatmEnt
Brief Title: Analysing Peripheral Skeletal Muscle Function Before and After Endobronchial Valve Treatment
Acronym: ENDURANCE
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Head of the department of Pulmonary Diseases and Pulmonologist, University Medical Center Groningen
Other Study IDs: ENDURANCE
Record Dates: First submitted 2023-08-04; First posted 2023-09-06 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle biopsies and peripheral blood collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EBV-patients: Patients who are scheduled for a bronchoscopic lung volume reduction treatment using endobronchial valves.
  Interventions: Diagnostic Test: 31P-Magnetic Resonance Spectroscopy (31P-MRS)

INTERVENTIONS:
Diagnostic Test: 31P-Magnetic Resonance Spectroscopy (31P-MRS) — 31P-Magnetic Resonance Spectroscopy will be performed during exercise testing.
  Other Names: Muscle biopsy

SUMMARY:
Rationale: Chronic obstructive pulmonary disease (COPD) is characterised by a high prevalence of peripheral muscle dysfunction, which can have significant clinical consequences, including decreased exercise capacity, reduced quality of life, and even a higher mortality rate. Reduction of lung hyperinflation using bronchoscopic lung volume reduction treatment with one-way endobronchial valves (EBV) is a minimally invasive intervention which improves exercise capacity and physical activity in patients with severe emphysema. This positive effect is also related to weight gain and alterations in body composition. The physiologic and structural adaptations of skeletal muscle function after EBV treatment has never been investigated before.

Objective: To investigate the physiological and structural adaptations of peripheral muscle function at a cellular level in response to EBV treatment.

Study design: A single center, prospective clinical trial with a single-arm pretest-posttest design. Patients with severe emphysema who will receive a bronchoscopic lung volume reduction treatment are asked to undergo additional in-magnet exercise testing and muscle biopsies before and after placement of EBVs.

Study population: Patients with severe emphysema who are scheduled to undergo EBV treatment.

Main study parameters/endpoints: The difference in quadriceps phosphocreatine concentration (PCr), quadriceps inorganic phosphorus concentration (Pi), and quadriceps pH at rest, during progressive exercise, and recovery rate will be measured by 31P-MRS to assess the physiological effect of EBV treatment on skeletal muscle function and its bioenergetics. Furthermore, we will perform a detailed histological and biochemical analysis of muscle fiber type composition, mitochondrial density, master regulators of muscle oxidative programming, and mitochondrial respiration before and after EBV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for a bronchoscopic lung volume treatment using one-way endobronchial valves;
* Patient read, understood and signed the Informed Consent Form.

Exclusion Criteria:

* Inability to perform a cycle ergometry test;
* Contraindications for undergoing a magnetic resonance imaging scan (e.g. claustrophobia, implanted cardiac devices);
* Body length >190cm;
* Any anticoagulant therapy;
* COPD exacerbation 4 weeks prior to testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population exists of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment with one-way endobronchial valves.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps phosphocreatine concentration measured by 31P-MRS. | 6 months
  To assess the physiological adaptations, in terms of cellular bioenergetics, of the quadriceps muscle in patients with severe COPD in response to EBV treatment. This will be done by performing 31P-MRS during exercise testing in a MR-compatible ergometer at baseline and at 6 months follow-up, for which the quadriceps phosphocreatine concentration (PCr) at rest and during progressive exercise will be assessed.

SECONDARY OUTCOMES:
Change in muscle fiber type composition measured in muscle biopsies. | 6 months
  Change in muscle fiber type composition 6 months after EBV treatment measured in muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — UMC Groningen
Locations (1):
- Univeristy Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on reasonable request